CLINICAL TRIAL: NCT05510752
Title: Cognitive Behavioural Therapy Versus Psychoeducation for Perinatal Anxiety: A Randomized Controlled Trial
Brief Title: Cognitive Behavioural Therapy Versus Psychoeducation for Perinatal Anxiety
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Sheryl Green, Associate Professor, Clinical Psychologist, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: CBT-Psychoed-RCT
Record Dates: First submitted 2022-08-15; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Perinatal Anxiety

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducation Group (Active Comparator): Psychoeducation is the most commonly offered non-pharmacological treatment for perinatal distress, with the assumption that an understanding of perinatal distress, self-care and infant milestones will improve mental health outcomes. Psychoeducation has been shown to be effective in reducing the severity of perinatal anxiety and depression.
  Interventions: Behavioral: Psychoeducation
- Cognitive Behavioural Group Therapy (Experimental): Cognitive Behavioural Group Therapy (CBGT) is a well-established psychological treatment for anxiety and other mental health disorders. CBGT treatment for perinatal anxiety has shown significant reductions in anxiety (primary outcome), worry and depression from pre- to post-treatment when compared to a waitlist control condition. However, to be considered well-established, a treatment must be at least as effective as other active interventions. As such, the present study will compare CBGT to what is most commonly offered to perinatal women with a principal anxiety disorder (i.e., psychoeducation).
  Interventions: Behavioral: Cognitive Behavioural Group Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioural Group Therapy — CBGT is a 6-week group that meets weekly for 2-hours per week, where participants learn cognitive and behavioural techniques to enhance coping skills for their everyday anxieties.
  Arms: Cognitive Behavioural Group Therapy
Behavioral: Psychoeducation — Psychoeducation is the most common non-pharmacological treatment for perinatal distress, where participants learn about healthy infant milestones and how to implement self-care in their daily lives, which in turn reduces distress during the perinatal period.
  Arms: Psychoeducation Group

SUMMARY:
Anxiety during pregnancy and the postpartum (perinatal) period is very common and is associated with adverse consequences for mothers and their infants. Currently, medication is the most commonly prescribed treatment for perinatal anxiety and the lack of nonmedication-based interventions for perinatal anxiety is a barrier to receiving effective treatment for many women. As such, the present single-blind, randomized controlled trial seeks to evaluate whether group-based cognitive behavioural therapy, the gold-standard psychological treatment for anxiety disorders in the general population, effectively treats perinatal anxiety symptoms when compared to a psychoeducation group, which is currently the most commonly prescribed non-medication-based treatment for perinatal distress.

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 and older that are pregnant or between 0-12 months postpartum;
2. Principal diagnosis of an anxiety disorder as per the Mini International Neuropsychiatric Interview for DSM-5 (version 7.0.2) with or without comorbid depression;
3. No concurrent psychological treatment;
4. Not taking psychoactive medication or a) medications are stable in dose and type for at least 8 weeks prior to the study (as per Canadian psychiatric guidelines; and b) medications remain stable throughout the study;
5. Fluent in English, minimal grade 8 reading level.

Exclusion Criteria:

1. Severe depression/suicidality requiring acute intervention;
2. Women with psychotic or current substance use disorders,
3. medication changes in dose or type or less than 5/6 sessions complete (will continue with treatment but be excluded from the study).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 216 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
State-Trait Inventory for Cognitive and Somatic Anxiety (STICSA) | Change from pre-treatment (baseline) to one week post-treatment to and 3-month follow up.
  The STICSA is a 21-item self-report scale that assesses cognitive and somatic components of anxiety. The STICSA is comprised of a state scale that measures individuals' current anxiety symptoms, and a trait scale that assesses one's proneness to anxiety, more generally. In the present study, only the trait scale of the STICSA will be used. Items are scored on a 4-point scale ranging from 1 ('not at all') to 4 ('very much so'). The STICSA has demonstrated excellent validity and reliability. A cut-off score of 43 or higher on the STICSA has been suggested for detecting a probable anxiety disorder. The STICSA has been validated for use in clinical samples of adults with anxiety disorders, although not explicitly in perinatal samples.

SECONDARY OUTCOMES:
Penn State Worry Questionnaire (PSWQ) | Change from pre-treatment (baseline) to one week post-treatment to and 3-month follow up.
  The PSWQ is a 16-item self-report measure that assesses the tendency to worry. Items are scored on a 5-point scale ranging from 1 ('not typical at all') to 5 ('very typical'), with higher scores reflecting greater pathological worry. A cut-off score of 62 or higher has been suggested for determining a probable GAD diagnosis. The PSWQ has demonstrated excellent internal consistency and validity across various populations and has been validated for use in perinatal samples.
Generalized Anxiety Disorder 7 (GAD-7) | Change from pre-treatment (baseline) to one week post-treatment to and 3-month follow up.
  The GAD-7 is a 7-item self-report measure that assesses anxiety symptom severity over a previous two-week period. Items are measured on a 4-point scale ranging from 0 ('not at all') to 3 ('nearly every day'). A cut-off score of 10 or higher with sensitivity of 89% and specificity of 82% has been suggested for detecting a probable diagnosis of Generalized Anxiety Disorder. The GAD-7 has also been validated for use in perinatal samples.
Edinburgh Postnatal Depression Scale (EPDS) | Change from pre-treatment (baseline) to one week post-treatment to and 3-month follow up.
  The EPDS is a 10-item self-report measure that assesses symptoms of depression during the perinatal period. Items are scored on a 4-point scale ranging from 0 to 3, with higher scores reflecting greater depressive symptomatology. The EPDS has demonstrated good sensitivity and specificity for a diagnosis of Major Depressive Disorder (MDD). Cut-off scores of 15 and 13 or higher have been suggested for detecting a probable diagnosis of MDD during pregnancy and the postpartum period, respectively.
Worry Behaviors Inventory Perinatal Revised (WBI-P) | Change from pre-treatment (baseline) to one week post-treatment to and 3-month follow up.
  The WBI-PR is adapted from the Worry Behaviours Inventory, which assesses the frequency of problematic behaviours associated with generalized anxiety disorder. The WBI-PR is a 10-item self-report measure that is designed to measure problematic GAD behaviours during the perinatal period. Items are measured on a 5-point Likert scale, ranging from 0 to 4 and includes two subscales: Avoidance and Safety Behaviours. In its initial validation, the WBI-PR demonstrated acceptable internal consistency and convergent and discriminant validity.
Intolerance of Uncertainty Scale (IUS) | Change from pre-treatment (baseline) to one week post-treatment to and 3-month follow up.
  The IUS is a 27-item self-report questionnaire assessing one's beliefs and reactions to uncertainty. Items are scored on a 5-point scale ranging from 1 ('not at all characteristic of me') to 5 ('entirely characteristic of me'), with higher scores reflecting greater intolerance of uncertainty. The IUS has demonstrated excellent internal consistency and test-retest reliability in the general population, and excellent convergent validity with measures of worry and GAD in perinatal populations. A cut-off score of 64 of greater with sensitivity of 89% and specificity of 65% has been determined for detection of an anxiety disorder within the perinatal period.
Perceived Stress Scale (PSS). | Change from pre-treatment (baseline) to one week post-treatment to and 3-month follow up.
  The PSS is the most widely used psychological instrument for measuring the perception of stress. The PSS is a 10-item self-report measure designed to assess the degree to which situations in one's life are appraised as stressful. Items are scored on a 5-point scale ranging from 0 ('never) to 4 ('fairly often') with higher scores reflecting greater perceived stress. The PSS has demonstrated good psychometric properties.
Difficulties in Emotion Regulation Scale (DERS) | Change from pre-treatment (baseline) to one week post-treatment to and 3-month follow up.
  The DERS is a 36-item self-report scale designed to assess difficulties with emotion regulation. The DERS contains six subscales that measure: non-acceptance goals, impulse, awareness, strategies, and clarity. Items are rated on a 5-point Likert scale, ranging from 1 (almost never, 0-10%) to 5 (almost always, 91-100%), with higher scores reflecting greater difficulties regulating emotions. The DERS has demonstrated good internal consistency (α=0.86) and test-retest reliability (0.74).
Insomnia Severity Index (ISI). | Change from pre-treatment (baseline) to one week post-treatment to and 3-month follow up.
  The ISI is a 7-item self-report questionnaire that assesses the nature, severity, and impact of insomnia. Items are scored on a 5-point Likert scale ranging from 0 ('no problem') to 4 ('very severe problem') with higher scores reflecting greater insomnia severity. Total scores between 0-7 indicate an absence of insomnia; scores between 8-14 suggest subthreshold insomnia; scores between 15-21 indicate moderate insomnia; and scores between 22-28 suggest severe insomnia. The ISI has demonstrated good psychometric properties.
Anxiety Sensitivity Index (ASI-3) | Change from pre-treatment (baseline) to one week post-treatment to and 3-month follow up.
  The ASI-3 is an 18-item self-report measures that assesses anxiety sensitivity related to physical, cognitive and social concerns. Items are scored on a 5-point scale ranging from 0 ('very little') to 4 ('very much'), with higher scores reflecting greater anxiety sensitivity. The ASI-3 has demonstrated good reliability and validity.
Abbreviated Dyadic Adjustment Scale (ADAS) | Change from pre-treatment (baseline) to one week post-treatment to and 3-month follow up.
  The ADAS is a 7-item self-report scale assessing relationship satisfaction and adjustment in couples. Six of the items are scored on a 6-point Likert Scale, with higher scores reflecting greater relationship satisfaction. Item seven provides a global 'overall happiness' rating and is scored on 7- point Likert Scale ranging from 0 (extremely unhappy) to 6 (perfect). The ADAS has demonstrated good internal consistency, validity, and responsivity to change.
Social Provisions Scale (SPS) | Change from pre-treatment (baseline) to one week post-treatment to and 3-month follow up.
  The SPS is a 24-item self-report scale that assesses perceived social support received within social relationships. Items are scored on a 4-point scale ranging from 1 (strongly disagree) to 4 (strongly agree), with higher scores indicating higher levels of perceived social support. The SPS has 6 subscales assessing dimensions of attachment, social integration, reassurance of worth, guidance, nurturance, and reliance.
Illness Intrusiveness Rating Scale (IIRS). | Change from pre-treatment (baseline) to one week post-treatment to and 3-month follow up.
  The IIRS is a 13-item self-report measure designed to assess the extent to which a particular problem causes impairment in different aspects of one's life including health, diet, work, recreation, finances, social and romantic relationships, sex life, self- and religious-expression, and community/civic involvement. Items are scores on a 7-point scale ranging from 1 ('not very much') to 7 ('very much'), with higher scores reflecting greater intrusiveness. The IIRS has shown good reliability and validity.
World Health Organization Quality of Life Scale (WHOQoL-BREF). | Change from pre-treatment (baseline) to one week post-treatment to and 3-month follow up.
  The WHOQoL-BREF is a 26-item self-report measure that assesses quality of life across four domains, including physical health, psychological health, social relationships, and environment (WHOQoL group, 1998). Items are scored on a 5-point Likert scale ranging from 1 to 5, with higher scores indicating greater quality of life. The WHOQoLBREF has demonstrated good discriminant validity, content validity, internal consistency, and test-retest reliability.
Client Satisfaction Questionnaire (CSQ) | One week post-treatment
  The CSQ is an 8-item self-report scale designed to measure satisfaction with health services. Items are scored on a 4-point scale from 1 to 4, with higher scores indicating higher levels of satisfaction with services. This scale demonstrates good psychometric properties with high internal consistency (Cronbach's alpha ranging from 0.92 to 0.93). In terms of construct validity, tests of global improvement correlated with client satisfaction (r = 0.53).

OTHER OUTCOMES:
Sociodemographic Factors | Change from pre-treatment (baseline) to one week post-treatment to and 3-month follow up.
  Sociodemographic information collected will include participant's gender, age, ethnicity, marital status, education level, income level, parity, medical and delivery history, family psychiatric history, medication usage, and treatment history.

IPD SHARING:
Plan to Share IPD: No